CLINICAL TRIAL: NCT03203681
Title: Natesto Effects on Testosterone, Luteinizing Hormone, Follicle Stimulating Hormone and Semen Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Director of Male Reproductive Medicine and Surgery/Assistant professor in Department of Urology at University of Miami, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170462
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Natesto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Natesto (Other): Participants in this group will receive Natesto for a 24 consecutive weeks treatment course.
  Interventions: Drug: Natesto

INTERVENTIONS:
Drug: Natesto — 4.5% nasal testosterone. 11.0 mg testosterone administered per dose (2 pump actuations, 1 pump per nostril) applied intranasally three times a day.

SUMMARY:
Low testosterone affects more than 10% of men worldwide, with high incidence in the elderly.This will be a prospective case study. The investigators will identify men with hypogonadism in our clinic interested in Natesto for testosterone replacement therapy (TRT). Natesto is a relatively new form of testosterone replacement therapy that is delivered intranasal to men diagnosed with low testosterone. Current advantages to Natesto include ease of delivery and decreased risk of transference. Recently Natesto 4.5% (125 uL/nostril, 11.0mg testosterone/dose), three times a day (TID) dosing was shown to also increase serum testosterone while maintaining normal, though decreased, serum levels of Luteinizing Hormone (LH) and Follicle-Stimulating Hormone(FSH). 40 participants will be enrolled and receive treatment with Natesto.The study will identify men with confirmed hypogonadism (testosterone (T) <350 on 2 consecutive Testosterone samples collected greater than 1.5 hours apart between 6am and 10am with demonstrated symptoms of hypogonadism). Participants with a history of prostate cancer, testis cancer, azoospermia, or genetic cause of hypogonadism will be excluded.

DETAILED DESCRIPTION:
Low testosterone affects more than 10% of men worldwide, with high incidence in the elderly). While Natesto has been shown to have positive effects on Testosterone while maintaining LH and FSH, the impact on sperm count has not yet been proven.

Study Design and Duration of Treatment: Participants will take Natesto 11g intra nasally there times a day (TID) for 16 weeks (120 days) between serum and semen evaluations.

Subject Population: The study will identify men with confirmed hypogonadism (testosterone (T) <350 on 2 consecutive Testosterone samples collected greater than 1.5 hours apart between 6am and 10am with demonstrated symptoms of hypogonadism). Subjects with a history of prostate cancer, testis cancer, azoospermia, or genetic cause of hypogonadism will be excluded.

Number of subjects: 40 participants will be enrolled and receive treatment with Natesto.

Study Duration:Total participation in the study will be approximately 24-28 weeks.

Study Procedures: Participants will undergo a total of six study visits. At the first visit, subjects will undergo screening procedures which will include signing of the consent form, physical exam, assessment for inclusion and exclusion criteria, Sexual Health Inventory in Men (SHIM) and quality of life questionnaire, blood sample for clinical laboratory assessment, and a semen analysis. At visit 2, subjects will undergo a second semen analysis and blood analysis for T. After 12 weeks (90 days), Participants will return for a third visit for blood sample and semen analysis as well as safety monitoring. The Participants will also be given SHIM and quality of life questionnaires. This procedure will be repeated at week 24 to get a final blood and semen analysis.

Study Endpoints: The primary endpoint will be change in FSH, LH, Estradiol, T, and Semen Analysis after 12 weeks and 24 weeks of treatment with Natesto. The secondary endpoint will be monitoring for adverse events

Statistical Methods: Analyses will consist of summaries of the values and total change from baseline in each value (visit value versus baseline value) using descriptive statistics (sample size, mean, median, standard deviation, 95% confidence interval, minimum, and maximum). The change from baseline in each endpoint will compared using a two-sample t-test, or the Wilcoxon rank sum test if distributional assumptions are violated. The primary time point of interest for assessing hormone effects is the week 12 visit.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign and date the study consent form(s) which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.
* Male between 18 and 55 years of age, inclusive, with documented onset of hypogonadism prior to age 55.
* Documented diagnosis of primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).
* Serum total testosterone < 350 ng/dL based on 2 consecutive blood samples obtained at least 1.5 hours apart between 6:00 am and 10:00 am following an appropriate washout of current androgen replacement therapy.
* Naïve to androgen replacement or has discontinued current treatment and completed a washout of 4 weeks following androgen treatment (excluding Testopel). Washout must be completed prior to collection of baseline serum testosterone samples to determine study eligibility.
* Judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of significant sensitivity or allergy to androgens, castor oil or product excipients.
* Clinically significant findings in the prestudy examinations including abnormal breast examination requiring follow-up, abnormal ECG.
* Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or International Prostate Symptoms Score (I-PSS) > 19 points.
* Body mass index (BMI) ≥ 30 kg/m2.
* Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

  1. Baseline hemoglobin < 11.5 g/dL or > 16 g/dL
  2. Hematocrit < 35% or > 54%
  3. Serum transaminases > 2.5 times upper limit of normal
  4. Serum bilirubin > 2.0 mg/dL
  5. Creatinine > 2.0 mg/dL f. Prostate-Specific Antigen (PSA) > 2 ng/mL
* History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
* History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration.
* History of stroke or myocardial infarction within the past 5 years.
* History of, or current or suspected, prostate or breast cancer.
* History of diagnosed, severe, untreated, obstructive sleep apnea.
* History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 12 weeks prior to the start of treatment.
* Inadequate venous access for collection of serial blood samples required for pharmacokinetic profiles.
* Receipt of any investigational product within 4 weeks or within 5 half-lives prior to the start of treatment.
* Inability to understand and provide written informed consent for the study.
* Considered by the investigator or the sponsor-designated physician, for any reason, that the subject is an unsuitable candidate to receive Natesto.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amory JK, Anawalt BD, Blaskovich PD, Gilchriest J, Nuwayser ES, Matsumoto AM. Testosterone release from a subcutaneous, biodegradable microcapsule formulation (Viatrel) in hypogonadal men. J Androl. 2002 Jan-Feb;23(1):84-91. doi: 10.1002/jand.2002.23.1.84. PMID 11780927
- [Background] Haring R, Ittermann T, Volzke H, Krebs A, Zygmunt M, Felix SB, Grabe HJ, Nauck M, Wallaschofski H. Prevalence, incidence and risk factors of testosterone deficiency in a population-based cohort of men: results from the study of health in Pomerania. Aging Male. 2010 Dec;13(4):247-57. doi: 10.3109/13685538.2010.487553. Epub 2010 May 26. PMID 20504090
- [Background] Kim ED, McCullough A, Kaminetsky J. Oral enclomiphene citrate raises testosterone and preserves sperm counts in obese hypogonadal men, unlike topical testosterone: restoration instead of replacement. BJU Int. 2016 Apr;117(4):677-85. doi: 10.1111/bju.13337. Epub 2015 Oct 23. PMID 26496621
- [Background] Ullah MI, Riche DM, Koch CA. Transdermal testosterone replacement therapy in men. Drug Des Devel Ther. 2014 Jan 9;8:101-12. doi: 10.2147/DDDT.S43475. eCollection 2014. PMID 24470750
- [Background] Rhoden EL, Morgentaler A. Risks of testosterone-replacement therapy and recommendations for monitoring. N Engl J Med. 2004 Jan 29;350(5):482-92. doi: 10.1056/NEJMra022251. No abstract available. PMID 14749457
- [Background] Rogol AD, Tkachenko N, Bryson N. Natesto , a novel testosterone nasal gel, normalizes androgen levels in hypogonadal men. Andrology. 2016 Jan;4(1):46-54. doi: 10.1111/andr.12137. Epub 2015 Dec 22. PMID 26695758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natesto
Started | 60
3 Month | 44
6 Months | 33
Completed | 33
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Natesto
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Demographics: Caucasian | 12
  Demographics: Black | 2
  Demographics: Hispanic | 34
  Demographics: Asian | 1
  Demographics: Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Testosterone Levels From Baseline to 27 Weeks
Description: Testosterone levels measured in ng/dL analyzed from peripheral venous puncture blood draw
Time Frame: Baseline, 27 Weeks
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Natesto
Number analyzed (Participants) | 33
ng/dL | 652 (305)

2. Primary Outcome: Change in Estradiol Levels From Baseline to 27 Weeks
Description: Estradiol levels measured in pg/mL analyzed from peripheral venous puncture blood draw
Time Frame: Baseline, 27 Weeks
Population: Estradiol levels were not collected for all participants that completed the study
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Natesto
Number analyzed (Participants) | 29
pg/mL | 21.6 (14)

3. Primary Outcome: Change in Gonadotropin Levels From Baseline to 27 Weeks
Description: Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) levels, both measured in mIU/mL analyzed from peripheral venous puncture blood draw
Time Frame: Baseline, 27 Weeks
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Natesto
Number analyzed (Participants) | 33
mIU/mL
  Follicle Stimulating Hormone | 3.0 (2.9)
  Luteinizing Hormone | 2.6 (3.1)

4. Primary Outcome: Number of Participants With an Increase in SF-36 QOL Scores From Baseline
Description: The number of participants with an increase of at least 1 point from their SF-36 QOL scores from baseline will be reported. Short Form-36 (SF-36) Quality of Life (QOL) questionnaire has a proprietary scoring system that ranges from 1-5 and each domain is individually assessed
Time Frame: 27 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Natesto
Number analyzed (Participants) | 33
Participants | 32

5. Primary Outcome: Change in Sperm Counts From Baseline to 27 Weeks
Description: Sperm count measured in million sperm/mL analyzed from semen sample
Time Frame: Baseline, 27 Weeks
Measure: Mean (Standard Deviation); unit: million sperm/mL
Arm/Group | Natesto
Number analyzed (Participants) | 33
million sperm/mL | 33.9 (24.3)

6. Primary Outcome: Incidence of Adverse Events
Description: Incidence of adverse events as assessed per treating physician
Time Frame: 27 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Natesto
Number analyzed (Participants) | 60
Participants
  Azoospermia | 1
  Severe Oligospermia | 3
  Nasal irritation | 5
  sinusitis | 1
  epistaxis | 1

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Natesto
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 4/60
Other Adverse Events (participants affected / at risk) | 5/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natesto (N=60)
Azoospermia (Reproductive system and breast disorders) | 1 (1)
Severe Oligospermia (Reproductive system and breast disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natesto (N=60)
Nasal Irritation (Injury, poisoning and procedural complications) | 5 (5)
Sinusitis (General disorders) | 1 (1)
Epistaxis (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03203681/Prot_SAP_000.pdf